CLINICAL TRIAL: NCT02699372
Title: A Single-center, Randomized, Investigator/Subject-Blind, Adaptive Single-ascending Dose (Part 1) and Multiple Ascending Dose (Part 2), Placebo-Controlled, Parallel Study to Investigate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of RO6889450 Following Oral Administration in Healthy Subjects
Brief Title: The Safety, Tolerability, Pharmacokinetics and Pharmacodynamics Study of RO6889450 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BP30134; 2015-005509-35 (EudraCT Number)
Record Dates: First submitted 2016-02-23; First posted 2016-03-04 (Estimated); Last update posted 2017-11-24 (Actual); Status verified 2017-11

CONDITIONS: Healthy Volunteer
Keywords: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- Placebo (Placebo Comparator): Healthy volunteers will receive the placebo equivalent to RO6889450 as oral capsules.
  Interventions: Drug: Placebo
- RO6889450: Part 1 Single Ascending Dose (SAD) (Experimental): Participants will undergo a series of screening visits prior to treatment and 4 weeks follow-up. Healthy volunteers will be enrolled in up to 7 dose groups (5 milligram [mg] to 450 mg) and will receive single oral dose of RO6889450 in the morning of the Day 1.
  Interventions: Drug: RO6889450
- RO6889450: Part 2 Multiple Ascending Dose (MAD) (Experimental): The starting dose for Part 2 MAD will be determined by analysis of safety and pharmacokinetic data of Part 1 SAD. All participants will receive RO6889450 orally for 14 days.
  Interventions: Drug: RO6889450

INTERVENTIONS:
Drug: Placebo
  Arms: Placebo
Drug: RO6889450
  Arms: RO6889450: Part 1 Single Ascending Dose (SAD); RO6889450: Part 2 Multiple Ascending Dose (MAD)

SUMMARY:
This randomized, single center, adaptive single ascending dose (Part 1) and multiple ascending dose (Part 2) study is designed to assess the safety, tolerability, pharmacokinetic, and pharmacodynamics following an oral administration of RO6889450 versus placebo in healthy volunteers. The anticipated duration of this study is approximately 18 weeks.

ELIGIBILITY:
Inclusion Criteria:

* A body mass index (BMI) between 18 to 30 kilogram per square meter (kg/m^2) inclusive
* Body weight in the range of 50 to 100 kilogram (kg) and right-handed - Part 2 only
* For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive methods
* For men: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive measures, and agreement to refrain from donating sperm
* Fluent in the language of the Investigator and study staff (including raters)
* Able to participate and comply with the study restrictions

Exclusion Criteria:

Part 1 and Part 2:

* Disorders of the central nervous system (CNS), psychiatric disorders, behavioral disturbances
* Participants who, in the Investigator's judgment, pose a suicidal or homicidal risk
* Any personal or familial history (first degree) of seizures, epilepsy or other convulsive condition
* Positive family history of psychosis or mood disorders up to first degree relative
* Angle closure glaucoma, history or current significant ophthalmologic or neurologic condition that would adversely affect the pupillometry assessment
* Suspicion of regular consumption of drug of abuse and/or any history of alcohol addiction with positive urine drug screen and/or positive alcohol urine test, or regular smoker
* Positive result on hepatitis B (HBV), hepatitis C (HCV), or human immunodeficiency virus antibody (HIV 1 and 2)
* Any prescribed or OTC medications (including vitamins or herbal remedies) taken within 4 weeks prior to first dosing or within 5 times the elimination half-life of the medication prior to first dosing (whichever is longer)
* Taking any nutrients known to modulate CYP3A activity (e.g., grapefruit juice; Seville orange) within 2 weeks prior to administration of study drugs
* Clinically significant abnormalities in laboratory test results (including hepatic and renal panels, complete blood count, chemistry panel and urinalysis)
* Participation in an investigational drug or device study within 90 days prior to screening
* Dietary restrictions that would prohibit the consumption of standardized meals
* Concomitant disease or condition that could interfere with, or treatment of which might interfere with, the conduct of the study, or that would, in the opinion of the investigator, pose an unacceptable risk to the participant in this study

Part 2:

* Contraindications for magnetic resonance imaging (MRI) scans or any brain/head abnormalities restricting MRI eligibility. Any sensorial impairment such as deafness and reduced visual acuity which cannot be corrected in the fMRI scanner
* Use of any psychoactive medication, or medications known to have effects on CNS or blood flow taken within 4 weeks prior to first dosing or within 5 times the elimination half-life of the medication prior to first dosing (whichever is longer)
* Fulfilment of any of the MRI contraindications on the standard radiography screening questionnaire

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 164 (Estimated)
Dates: Start 2016-03-21 (Actual); Primary Completion 2017-04-14 (Actual); Study Completion 2017-04-14 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants With Dose Limiting Toxicities After Single Ascending Dose (SAD) - Part 1 | up to 22 days
Area Under the Curve from Time Zero to end of dosing interval (AUCtau) After Multiple Oral Ascending Doses - Part 2 | Part 2: predose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16 hr postdose on Day 1; predose on Days 2, 3, 4, 5, 6, 7, 8, 10, 12, 13, predose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16 hr postdose on Day 14, Days 15, 16, 17, 19, 20, 21
Percentage of Participants With Dose Limiting Toxicities After Multiple Oral Ascending Doses (MAD) - Part 2 | up to 35 days
Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC (0 to inf)] After Single Ascending Dose - Part 1 | Part 1: predose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16 hours (hr) postdose on Day 1; Day 2, 3, 4, 6, 7, 8
RO6889450 Maximum Plasma Concentration (Cmax) After Single Oral Ascending Doses | Part 1: predose and 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16 hours postdose on Day 1, Days 2, 3, 4, 6, 7, 8
RO6889450 Maximum Plasma Concentration (Cmax) After Multiple Oral Ascending Doses | Part 2: predose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16 hours postdose on Day 1, predose on Days 2, 3, 4, 5, 6, 7, 8, 10, 12, 13, predose and 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16 hours postdose on Day 14, Days 15, 16, 17, 19, 20, 21
RO6889450 Minimum Observed Plasma Trough Concentration (Cmin) | Part 2: predose on Days 2, 3, 4, 5, 6, 7, 8, 10, 12, 13, predose and 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16 hours postdose on Day 14, Days 15

SECONDARY OUTCOMES:
Time to Reach Maximum Observed Plasma Concentration (Tmax) After Multiple Ascending Dose - Part 2 | predose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16 hr postdose, Days 2, 3, 4, 5, 6, 7, 8, 10, 12, 13, predose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16 hr postdose on Day 14, Days 15, 16, 17, 19, 20, 21
Terminal Rate Constant After Multiple Ascending Dose - Part 2 | Part 2: predose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16 hr postdose on Day 1, predose on Days 2, 3, 4, 5, 6, 7, 8, 10, 12, 13, predose, 0.5,1,1.5, 2, 2.5, 3,4, 6, 8, 12, 16 hr postdose on Day 14, Days 15, 16, 17, 19, 20, 21
Apparent Terminal Half-Life (t1/2) After Multiple Ascending Dose - Part 2 | Part 2: predose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16 hr postdose on Day 1, predose on Days 2, 3, 4, 5, 6, 7, 8, 10, 12, 13, predose, 0.5, 1, 1.5, 2, 2.5, 3,4, 6, 8, 12, 16 hr postdose on Day 14, Days 15, 16, 17, 19, 20, 21
Apparent Oral Clearance (CL/F) After Multiple Ascending Dose - Part 2 | Part 2: predose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16 hr postdose on Day 1, predose on Days 2, 3, 4, 5, 6, 7, 8, 10, 12, 13, predose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16 hr postdose on Day 14, Days 15, 16, 17, 19, 20, 21
Cumulative Amount Excreted Unchanged in Urine (Ae) After Multiple Ascending Dose - Part 2 | Part 2: predose, 0 to 6, 6 to 12, 12 to 24 hours postdose on Day 1, 14, 24 to 48 and 48 to 72 hours after Day 14 dosing
Renal Clearance (CLR) After Multiple Ascending Dose - Part 2 | Part 2: predose, 0 to 6, 6 to 12, 12 to 24 hours postdose on Day 1, 14, 24 to 48 and 48 to 72 hours after Day 14 dosing
Fasting Glucose Concentrations After Multiple Ascending Dose - Part 2 | Part 2: Baseline, Days 7, 15, 17
Plasma Concentration of Prolactin - Part 2 | Part 2: Day 1, 14, 15
Scotopic Pupil Diameter as Assessed by Pupillometer - Part 2 | Part 2: Day 1, 2, 14, 15
Time to Reach Maximum Observed Plasma Concentration (Tmax) After Single Ascending Dose - Part 1 | Part 1: predose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16 hours (hr) postdose on Day 1, Days 2, 3, 4, 6, 7, 8
Last Measurable Concentration (Clast) After Single Ascending Dose - Part 1 | Part 1: predose and 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16 hours postdose on Day 1, Days 2, 3, 4, 6, 7, 8
Time to Last Measurable Concentration (Tlast) After Single Ascending Dose - Part 1 | Part 1: predose and 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16 hours postdose on Day 1, Days 2, 3, 4, 6, 7, 8
Terminal Rate Constant After Single Ascending Dose - Part 1 | Part 1: predose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16 hr postdose on Day 1, Days 2, 3, 4, 6, 7, 8
Apparent Terminal Half-Life (t1/2) After Single Ascending Dose - Part 1 | Part 1: predose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16 hr postdose on Day 1, Days 2, 3, 4, 6, 7, 8
Area Under the Plasma Concentration Versus Time Curve From Zero to 24 Hours Post-Dose (AUC0-24h) After Single Ascending Dose - Part 1 | Part 1: predose and 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16 hours postdose on Day 1, Days 2, 3, 4, 6, 7, 8
Area Under the Plasma Concentration Versus Time Curve up to the Last Measurable Concentration (AUC0-last) After Single Ascending Dose - Part 1 | Part 1: predose and 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16 hours postdose on Day 1, Days 2, 3, 4, 6, 7, 8
Apparent Oral Clearance (CL/F) After Single Ascending Dose - Part 1 | Part 1: predose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16 hr postdose on Day 1, Days 2, 3, 4, 6, 7, 8
Cumulative Amount Excreted Unchanged in the Urine (Ae) After Single Ascending Dose - Part 1 | Part 1: predose, 0 to 6, 6 to 12, 12 to 24 hours postdose on Day 1, 24 to 48, 48 to 72 hours after Day 1 dosing
Renal Clearance (CLR) After Single Ascending Dose - Part 1 | Part 1: predose, 0 to 6, 6 to 12, 12 to 24 hours postdose on Day 1, 24 to 48, 48 to 72 hours after Day 1 dosing
Accumulation Ratio for AUCtau (RAUC), Calculated as Day 14 AUC0-tau/Day 1 AUC0-tau - Part 2 | predose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16, 24 hours (hr) postdose on Day 1; predose, 0.5,1,1.5, 2, 2.5, 3,4, 6, 8, 12, 16, 24 hr postdose on Day 14
Accumulation Ratio for Cmax (RCmax), Calculated as Day 14 Cmax / Day 1 Cmax - Part 2 | predose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16 hours (hr) postdose on Day 1; predose, 0.5,1,1.5, 2, 2.5, 3,4, 6, 8, 12, 16, 24 hr postdose on Day 14
Accumulation Ratio for Ctrough RCtrough, Calculated as Day 14 Ctrough / Day 1 Ctrough - Part 2 | predose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16 hours (hr) postdose on Day 1; predose, 0.5,1,1.5, 2, 2.5, 3,4, 6, 8, 12, 16, 24 hr postdose on Day 14
Fasting Glucose Concentrations After Single - Part 1 | Part 1: Baseline, Day 4
Change From Baseline in Glucose Level at Day 14 - Part 2 | Baseline, Day 14
Change From Baseline in Insulin Level at Day 14 - Part 2 | Baseline, Day 14
Change From Baseline in C-peptide Level at Day 14 - Part 2 | Baseline, Day 14
Change From Baseline in Gastric Inhibitory Polypeptide (GIP) Level at Day 14 - Part 2 | Baseline, Day 14
Change From Baseline in Glucagon-like Peptide-1 (GLP-1) Level at Day 14 - Part 2 | Baseline, Day 14
Columbia Suicide-Severity Rating Scale (C-SSRS) Scores - Part 1 | Part 1: Day 4
Columbia Suicide-Severity Rating Scale (C-SSRS) Scores - Part 2 | Part 2: Day 15
Capillary Blood Glucose Levels - Part 1 | Part 1: Baseline through Day 4
Capillary Blood Glucose Levels - Part 2 | Part 2: Baseline through Day 17
Urine Concentration of Dopamine Metabolite - Part 2 | Baseline, Day 12, Day 13
Plasma Concentration of Prolactin - Part 1 | Part 1: Day 1, Day 2
Change From Baseline in Body Weight at Days 7 and 15 - Part 2 | Baseline, Day 7, 15
Addiction Research Center Inventory (ARCI-49) Questionnaire Score - Part 2 | Baseline, Day 1, 7, 14
Scotopic Pupil Diameter as Assessed by Pupillometer - Part 1 | Part 1: Day 1, 2
Change From Baseline in Regional Cerebral Blood Flow (CBF), as Assessed by Functional Magnetic Resonance Imaging (fMRI) at Days 7 or 8, 12 or 13 | Baseline, Day 7 or 8, 12 or 13
Facial Expression Recognition Task (FERT) Score, as Assessed by Emotional Test Battery (ETB) - Part 2 | Baseline, Day 12 or 13
Reward Learning Task Score, as Assessed by Effort-Based Paradigms - Part 2 | Baseline, Day 12 or 13

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- PRA Health Sciences Early Development Services, Zuidlaren, Netherlands